CLINICAL TRIAL: NCT02730884
Title: A Phase II Single-Arm Study of the Efficacy and Safety of Oral Rigosertib in Patients With Myelofibrosis (MF) and Anemia
Brief Title: Single-Arm Study of the Efficacy and Safety of Oral Rigosertib in Patients With Myelofibrosis (MF) and Anemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated Per PIs request due to low accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0546; NCI-2016-00761 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2016-03-24; First posted 2016-04-07 (Estimated); Results first posted 2020-08-07 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Leukemia; Myelofibrosis; Anemia; Splenomegaly
Keywords: Leukemia; Myelofibrosis; MF; Anemia; Splenomegaly; Post-polycythemia vera MF; post-PV; post-essential thrombocythemia MF; post-ET; Rigosertib; ON 01910.Na; Questionnaire; Survey
MeSH Terms: conditions — Leukemia; Primary Myelofibrosis; Anemia; Splenomegaly | interventions — ON 01910; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rigosertib (Experimental): Participants receive oral Rigosertib under fasting conditions twice a day on a continuous basis. Quality of life questionnaire completed on Day 1 of Cycle 1.
  Interventions: Drug: Rigosertib; Behavioral: Questionnaire

INTERVENTIONS:
Drug: Rigosertib — Participants take 560 mg Rigosertib by mouth in the morning (two 280 mg capsules) and 560 mg Rigosertib in the afternoon.
  Other Names: ON 01910.Na
Behavioral: Questionnaire — Quality of life questionnaire completed on Day 1 of Cycle 1. It should take about 10-15 minutes to complete.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is to learn if rigosertib can help to control MF in patients with anemia. The safety of this drug will also be studied.

This is an investigational study. Rigosertib is not FDA-approved or commercially available. It is currently being used for research purposes only. The study doctor can explain how the study drug is designed to work.

Up to 35 participants will be enrolled in this study. All will be enrolled at MD Anderson.

DETAILED DESCRIPTION:
Study Drug Administration:

If participant is found to be eligible to take part in this study, participant will take rigosertib capsules by mouth 2 times each day (1 morning dose, 1 afternoon dose) for 48 weeks. Participant will take participant's morning dose on an empty stomach. Participant's afternoon dose should be taken at about 3:00 pm (±1 hour), at least 2 hours after lunch. Participant should drink at least a ½ gallon of water each day. Rigosertib should be refrigerated.

Participant will also be given a study drug diary. Participant should write down each dose of study drug that participant takes, when participant takes it, and if participant misses or vomit any doses. If participant misses or vomits a dose of rigosertib, participant should not make up the dose. Participant should take the next scheduled dose as planned. Every 4 weeks for 12 weeks, then every 8 weeks thereafter, participant should bring any leftover rigosertib capsules and participant's study drug diary with participant to the clinic.

Study Visits:

On Cycle 1 Day 1:

* Participant will have a physical exam.
* Blood (about 2-3 teaspoons) and urine will be collected for routine tests.
* Blood (about 2 teaspoons) will be drawn for pharmacokinetic (PK) testing about 1 hour after participant's dose of study drug. PK testing measures the amount of study drug in the body at different time points.
* Participant will complete a questionnaire about participant's quality of life. It should take about 10-15 minutes.
* If the doctor thinks it is needed, participant will have a computed tomography (CT) or magnetic resonance imaging (MRI) scan to check the status of the disease.

Each week, blood (about 2-3 teaspoons) will be drawn for routine tests. If the study doctor approves it, participant may have these weekly blood draws at a local lab closer to participant's home. The results from these routine tests will be sent to the study doctor.

On Day 1 of Week 4, blood (about 2 teaspoons each time) will be drawn for PK testing before and 1 hour after participant's dose of study drug.

At Weeks 24 and 48 (± 1 week):

* Participant will have a bone marrow aspirate/biopsy performed to check the status of the disease. This sample may also be used for cytogenetic testing.
* If participant had a CT/MRI scan performed during Week 1, participant will have another CT/MRI scan to check the status of the disease.
* If participant can become pregnant, urine will be collected for a pregnancy test.

Every 4 weeks until Week 12 and then every 8 weeks after that:

* Participant will have a physical exam.
* Blood (about 2-3 teaspoons) and urine will be collected for routine tests.
* Participant will complete a questionnaire about participant's quality of life.

Length of Study:

Participant may continue taking the study drug for up to 48 weeks. Participant will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if participant is unable to follow study directions.

If the doctor thinks it is in participant's best interest, participant may be able to continue taking the study drug after 48 weeks. The study doctor will discuss this with participant.

Participation on the study will be over after the end-of-study visit.

End-of-Study Visit:

About 4 weeks after participant's last dose of study drug, participant will have an end-of-study visit. At this visit:

* Participant will have a physical exam.
* Blood (about 2-3 teaspoons) and urine will be collected for routine tests. This routine blood and urine collection will also include a pregnancy test if participant can become pregnant.

ELIGIBILITY:
Inclusion Criteria:

1. >/= 18 years of age;
2. Diagnosis of primary myelofibrosis (PMF) or post-polycythemia vera (post-PV) MF or post-essential thrombocythemia (post-ET) MF based on the World Health Organization (WHO) criteria or the International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT) criteria, which must be confirmed by BM aspirate and/or biopsy within 6 weeks prior to Screening. Measurement of JAK2 V617F allele burden in Bone Marrow (BM) samples, if not done within 6 months prior to Screening, must be provided with the Screening BM biopsy/aspirate report (patients are eligible regardless of JAK2 mutation status);
3. Anemia or RBC-transfusion dependence defined as follows: a) Anemia: defined for the purpose of this protocol as 1) a hemoglobin level <10 g/L on every determination over 84 days before study-entry, without red blood cell (RBC)-transfusions, or 2) a hemoglobin level <10 g/L on a patient that is receiving RBC-transfusions periodically but not meeting criteria for transfusion-dependent patient as defined below. The baseline hemoglobin value for these subjects is the lowest hemoglobin level during the antecedent 84 days; b) RBC-transfusion-dependence: RBC-transfusion-frequency of >/=2 units packed red blood cells (PRBC)/28 days averaged over 84 days immediately pre-study-entry. There must not be any consecutive 42 days without an RBC-transfusion during this interval.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2;
5. Willing to adhere to the prohibitions and restrictions specified in this protocol (Notation: the subject's willingness to adhere to prohibitions and restrictions must be clearly communicated in the on-study note);
6. The patient must signed an informed consent form (ICF) indicating that s/he understands the purpose of, and procedures required for, the study and is willing to participate.

Exclusion Criteria:

1. Ongoing clinically significant anemia due to factors such as known iron, vitamin B12, or folate deficiencies, auto-immune or hereditary hemolysis, or gastrointestinal (GI) bleeding;
2. Serum ferritin < 50 ng/mL;
3. Any active malignancy within the past year, except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix or breast; patients with history of prior malignancies should be free of disease for at least 3 years to be eligible for this study.
4. Uncontrolled intercurrent illness, including, but not limited to symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia;
5. Active infection not adequately responding to appropriate therapy;
6. Direct bilirubin >/= 2.0 mg/dL not related to hemolysis or Gilbert's disease;
7. Alanine transaminase (ALT) or aspartate transaminase (AST)>/= 2.5 x the upper limit of normal (ULN);
8. Serum creatinine >/= 2.5 mg/dL;
9. Ascites requiring active medical management including paracentesis;
10. Hyponatremia (defined as serum sodium level < 130 mEq/L);
11. Female patients who are pregnant or lactating;
12. Patients of childbearing potential (ie, women of childbearing potential and men with female partners of childbearing potential) who are unwilling to follow strict contraception requirements (including 2 reliable methods in combination: 1 non-hormonal, highly-reliable method [diaphragm, condoms with spermicidal foam or jelly, or sterilization] plus 1 additional reliable method [birth control pills, intrauterine device, contraceptive injections, or contraceptive patches]) before entry and throughout the study, up to and including the 30-day non-treatment follow-up period;
13. Female patients of childbearing potential who have a positive blood or urine pregnancy test at Screening;
14. Major surgery without full recovery or major surgery within 3 weeks of Screening;
15. Uncontrolled hypertension (defined as a sustained systolic pressure >/= 160 mmHg and/or a diastolic pressure >/= 110 mmHg);
16. New onset seizures (within 3 months prior to Screening) or poorly controlled seizures;
17. Any other concurrent investigational agent or chemotherapy, radiotherapy, or immunotherapy;
18. Chronic use (> 2 weeks) of corticosteroids (prednisone >/= 10 mg/24 hr equivalent) within 4 weeks of Screening;
19. Investigational therapy within 2 weeks of Screening;
20. Psychiatric illness or social situation that would limit the patient's ability to tolerate and/or comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: August 2017 to April 2019
Period: Overall Study
Arm/Group | Rigosertib
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rigosertib
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 67 [59 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Spleen Volume Response
Description: Spleen response defined as ≥ 35% spleen volume reduction from Baseline, which must be confirmed by MRI or CT measurement per revised International Working Group for Myelofibrosis Research and Treatment (IWG MRT) response criteria.
Time Frame: Baseline and 48 weeks
Population: of the three participants, one participant was not evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Rigosertib
Number analyzed (Participants) | 2
Participants | 0

2. Primary Outcome: Participants With Anemia Response
Description: Anemia response defined as the proportion of transfusion-independent patients with Hgb increase of at least 2 g/dL from Baseline or the proportion of transfusion-dependent patients becoming transfusion independent for at least 12 weeks as defined in 2013 International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) criteria.
Time Frame: Baseline and 48 weeks
Population: of the three participants, one participant was not evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Rigosertib
Number analyzed (Participants) | 2
Participants | 0

3. Secondary Outcome: Symptoms Response
Description: Symptoms response defined as the proportion of patients achieving ≥ 50% reduction in the Myeloproliferative Neoplasm Symptom Assessment Form Total Symptom Score (MPN-SAF TSS) at any time before Week 48.
Time Frame: 48 weeks
Population: of the three participants, one participant was not evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Rigosertib
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Rigosertib
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rigosertib (N=3)
Anemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rigosertib (N=3)
Neutrophil Count Decrease (Investigations) | 1 (1)
Would Infection (Infections and infestations) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombocytopenia (Investigations) | 1 (1)
Dirrhea (Gastrointestinal disorders) | 1 (1)
Acute Congestive Heart Failure (Cardiac disorders) | 1 (1)
Urinary Tract Pain (Renal and urinary disorders) | 1 (1)
Gastroparesis (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/84/NCT02730884/Prot_SAP_000.pdf